CLINICAL TRIAL: NCT05393531
Title: Comparison of First Line Non-invasive Treatment Options in Patients Diagnosed With Obstructive Sleep Apnea
Brief Title: First Line Obstructive Sleep Apnea Treatment Study
Acronym: FLOSAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: B300202100205
Record Dates: First submitted 2021-11-24; First posted 2022-05-26 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Mandibular Advancement Device; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints; Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mandibular advancement device (Other): Active therapy
  Interventions: Device: Mandibular advancement device (MAD)
- Continuous positive airway pressure (Other): Active therapy
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Mandibular advancement device (MAD) — Active therapy
  Other Names: EVO Prosomnus
  Arms: Mandibular advancement device
Device: Continuous positive airway pressure (CPAP) — Active therapy
  Other Names: Philips Respironics - Dreamstation
  Arms: Continuous positive airway pressure

SUMMARY:
The main objective is to evaluate the overall effectiveness of MAD therapy as a first line treatment, including both efficacy in terms of reduction in OSA severity as well as objective compliance, in patients recently diagnosed with moderate to severe OSA, waiting for a new CPAP device.

Upon completion of MAD-therapy, patients will be put on CPAP, allowing for comparison of MAD effectiveness versus the overall therapeutic effectiveness of CPAP therapy in the same patient.

Finally, patients' preference for either therapy will be evaluated.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent disorder, affecting up to 17% of middle-aged men. OSA is characterized by repetitive narrowing (hypopnea) or complete collapse (apnea) of the upper airway during sleep. This can cause intermittent breathing cessation during sleep, which leads to oxygen desaturation and micro-arousals during the night and eventually sleep fragmentation. Due to these perturbations, OSA is linked to a range of harmful sequelae: excessive daytime sleepiness, fatigue, an impaired cognitive performance, a reduced quality of life, an increased risk of occupational and traffic accidents, metabolic disturbances, hypertension, cardio- and cerebrovascular morbidity and OSA-related mortality. OSA severity is characterized by the apnea-hypopnea index (AHI), representing the amount of apneas and hypopneas during at least ten seconds, per hour of sleep. When studying OSA, one can also use the obstructive apnea-hypopnea index (OAHI) leaving out any central apnea component.

Due to the high prevalence as well as the individual and socioeconomic healthcare issues related to OSA, effective management of this chronic disorder is imperative. Continuous positive airway pressure (CPAP) is typically recommended as first line therapy for moderate to severe OSA, applying pressurized air throughout the respiratory cycle to keep the upper airway patent. Although CPAP is highly efficacious in reducing the severity of OSA, the clinical effectiveness is often compromised by a low patient acceptance and suboptimal adherence.

The alternative non-invasive treatment option is the use of a mandibular advancement device (MAD): this type of oral appliance protrudes the mandible during sleep, thereby enlarging and stabilizing the upper airway. The efficacy of MAD therapy in terms of reduction in AHI is demonstrated in clinical trials but turns out to be less efficacious compared to that obtained with CPAP. However, this suboptimal efficacy is counterbalanced by a higher compliance rate and relatively low discontinuation rate.

Nevertheless, studies comparing MAD with CPAP therapy outcomes show that both therapies are equally effective in reducing blood pressure and in reducing cardiovascular death. This might be explained by the greater efficacy of CPAP being offset by inferior compliance relative to MAD, resulting in similar clinical effectiveness. However, such studies are generally lacking objective compliance measurements for MAD therapy.

At this moment, different models of CPAP machines made by Philips Respironics were recalled in June 2021 due to a potential health risk: the polyester-based polyurethane sound abatement foam, which is used to reduce sound and vibration in these affected devices, may break down and potentially enter the device's air pathway. If this occurs, black debris from the foam or certain chemicals released into the device's air pathway may be inhaled or swallowed by the patient using the device. This indirectly implicates that there is a supply chain problem regarding new CPAP devices for patients recently diagnosed with moderate to severe OSA, and that those patients stay untreated until this supply chain problem is resolved. Up till now, this time frame is unclear.

Study protocol The investigators will perform a crossover clinical trial comparing the overall effectiveness of MAD therapy with the effectiveness of CPAP therapy in terms of reduction in OAHI.

The investigators will include patients that are diagnosed with moderate to severe OSA (obstructive AHI ≥ 15 events/hour of sleep and < 65 events/hour of sleep), body mass index < 35 kg/m² and put on the waiting list to receive CPAP therapy but that underwent the CPAP titration night.

Those patients will be invited to start MAD therapy with a custom-made titratable MAD (ProSomnus EVO, ProSomnus, Pleasanton, CA, USA). The MAD devices will be provided free of charge and an active thermomicrosensor (Theramon, IFT Handels- und Entwicklungsgesellschaft GmbH, Handelsagentur Gschladt) will be embedded to objectively measure the adherence to MAD therapy. The patients are then treated according to routine clinical practice: after three months of MAD use, the efficacy of the therapy in terms of reduction in OSA severity will be evaluated in the real life setting by using a portable home sleep test. The objective adherence will be read out from the thermomicrosensor, in order to be able to calculate the overall clinical effectiveness of this given therapy.

After this objective evaluation of the clinical effectiveness of MAD therapy, a wash-out period of one week is integrated in the protocol. Thereafter, when CPAP devices are available again and at least three months after the start of MAD therapy, patients will start with CPAP therapy. After three months of CPAP use, the efficacy in terms of reduction in OSA severity will be evaluated in the real life setting by using a portable home sleep test. Also, the objective adherence will be read out using the built-in registration data, to calculate the overall clinical effectiveness.

At the end of the study, patients will be questioned regarding their treatment preference: do they prefer CPAP, MAD or do they have no preference at all.

ELIGIBILITY:
Inclusion Criteria:

* oAHI ≥ 15 events/hour of sleep and < 65 events/hour of sleep
* BMI < 35 kg/m²
* waiting list to receive CPAP therapy but underwent the CPAP titration night

Exclusion Criteria:

* dental status not good enough for MAD therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Overall therapeutic effectiveness of MAD and CPAP | 3 months after start of the therapy (either MAD or CPAP)
  Combination of adherence (hours use per night) and efficacy (decrease in apnea/hypopnea index measured during a polysomnography)

SECONDARY OUTCOMES:
Treatment preference by questionnarie: which treatment do you prefer: CPAP, MAD or none? | 6 months
  Preference of the patients for one of the two given therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No